CLINICAL TRIAL: NCT07339215
Title: A Prospective Randomized Trial of Local Antibiotic Carriers in Tissue Expander-Based Breast Reconstruction
Brief Title: Local Antibiotic Concentrations With Tissue Expanders in Breast Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2369088
Record Dates: First submitted 2025-12-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Tissue Expander Based Breast Reconstruction
Keywords: breast reconstruction; Tissue Expander Breast Reconstruction; Tissue Expander; Surgical Site Infection; Periprosthetic Infection; Local antibiotics; PMMA antibiotic disc
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either an antibiotic-impregnated PMMA disc or absorbable antibiotic beads placed in the breast pocket at the time of tissue expander reconstruction. Each participant remains in their assigned group for the duration of the study, with no crossover between arms.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PMMA Antibiotic Disc (Experimental): Participants in this arm will receive a non-absorbable PMMA disc containing vancomycin and tobramycin placed in the breast pocket at the time of tissue expander reconstruction.
  Interventions: Device: Polymethylmethacrylate antibiotic disc
- Absorbable Antibiotic Beads (Active Comparator): Participants in this arm will receive absorbable antibiotic beads containing vancomycin and tobramycin placed in the breast pocket at the time of tissue expander reconstruction.
  Interventions: Device: Antibiotic loaded calcium sulfate beads

INTERVENTIONS:
Device: Antibiotic loaded calcium sulfate beads — Absorbable antibiotic beads containing vancomycin and tobramycin will be placed in the breast pocket at the time of tissue expander reconstruction. The beads dissolve gradually and release antibiotics directly into the periprosthetic space. This intervention allows comparison of antibiotic exposure, infection rates, and tissue expander complications relative to the non-absorbable PMMA disc.
  Arms: Absorbable Antibiotic Beads
Device: Polymethylmethacrylate antibiotic disc — A non-absorbable polymethylmethacrylate (PMMA) disc containing vancomycin and tobramycin will be placed in the breast pocket at the time of tissue expander reconstruction. The disc is molded intraoperatively and designed to elute high local concentrations of antibiotics into the periprosthetic space. This intervention is intended to reduce early postoperative infection risk and allow pharmacokinetic sampling of antibiotic levels in seroma fluid during routine postoperative visits.
  Arms: PMMA Antibiotic Disc

SUMMARY:
Infections after tissue expander breast reconstruction can lead to pain, additional surgeries, and loss of the reconstruction. This study will compare two types of antibiotic carriers used during surgery to help lower the risk of infection. One carrier is a non-absorbable PMMA disc, and the other is an absorbable antibiotic bead. Both release antibiotics directly into the breast pocket after surgery.

About 100 patients will be randomly assigned to receive one of these two carriers at the time of tissue expander placement. After surgery, small samples of fluid around the tissue expander will be collected during routine clinic visits. These samples will be tested to measure how much antibiotic is present over time. The study will also track infections, tissue expander loss, and other complications during the first 90 days after surgery. The goal is to learn how much antibiotic each carrier delivers and whether one method is more effective at preventing infection.

DETAILED DESCRIPTION:
Infection remains a devastating complication in tissue expander-based breast reconstruction, potentially causing patient distress, multiple re-operations, explantation, and the failure of the entire reconstructive process. A promising strategy to reduce this risk involves the local application of antibiotic carriers-materials placed in the surgical pocket that elute high concentrations of antibiotics directly at the site where infections begin. Recent studies have shown that both non-absorbable polymethylmethacrylate (PMMA) discs and absorbable antibiotic beads can significantly lower infection rates. However, the current evidence is limited because all prior studies are retrospective, lack direct comparisons between these carriers, and crucially, have no measurements of the actual antibiotic levels achieved in patients. This gap in knowledge leaves surgeons without clear, evidence-based guidance on which method is superior. This study is a prospective, randomized controlled trial designed to provide that definitive evidence. The investigators will enroll 100 patients undergoing tissue expander breast reconstruction at our institution. During surgery, each participant will be randomly assigned to receive either an antibiotic-impregnated PMMA disc or absorbable antibiotic beads placed in the breast pocket alongside the tissue expander. The study is meticulously designed to eliminate bias, with independent experts blinded to the treatment when assessing outcomes. The primary objective is to conduct a detailed pharmacokinetic analysis, measuring the concentration of vancomycin and tobramycin in the periprosthetic fluid over time. This will be achieved by analyzing seroma fluid aspirated during routine, scheduled post-operative clinic visits. This novel approach will not only provide data on whether the carriers work, but also how they work-how high the antibiotic levels reach, and for how long they remain effective. The secondary objective is to compare critical clinical outcomes, including surgical site infection rates, tissue expander loss, and other complications over a 90-day period. By directly linking precise, local drug exposure data with hard clinical endpoints, this research will for the first time establish a biologic gradient for efficacy and determine the comparative effectiveness of these two infection-prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females ≥18 years undergoing TE-based breast reconstruction (immediate or delayed).
2. Able to consent and comply with follow-up/aspiration visits.

Exclusion Criteria:

1. Allergy to vancomycin, tobramycin, or PMMA components.
2. CKD stage 4-5 (eGFR <30 mL/min/1.73m²).
3. Chronic immunosuppression (≥10 mg prednisone daily or biologic immunosuppressants).
4. Active systemic infection
5. Pregnancy, planning to become pregnant during the study, or lactation.
6. Lack of capacity to provide consent.
7. Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Local antibiotic exposure (log-transformed AUC₀-₄ weeks) | Perioperative/Periprocedural
  Vancomycin and tobramycin concentrations will be measured in periprosthetic seroma fluid collected during routine postoperative visits. The primary endpoint is the log-transformed area under the concentration-time curve from week 0 to week 4 (AUC₀-₄ weeks), which will be compared between the PMMA disc and absorbable bead groups. This will be measured weekly from tissue expander placement (baseline), and weekly at each tissue expander fill until tissue expander exchange at 4 weeks.

SECONDARY OUTCOMES:
Surgical site infection rate | Perioperative/Periprocedural
  Infections will be defined using CDC criteria. A blinded adjudication committee will review all suspected cases. The incidence of infection within 90 days after tissue expander placement will be compared between arms.
Tissue expander loss | Perioperative/Periprocedural
  Tissue expander loss is defined as explantation due to infection, wound breakdown, or other complications. The proportion of patients requiring explantation within 90 days of surgery will be compared between groups.
Peak antibiotic concentration (Cmax) | Perioperative/Periprocedural
  Antibiotic concentrations of aspirated Seroma fluid will be measured at the time of tissue expander placement (baseline), and weekly there-after at the time of tissue expander fills from week 1 to week 4. The highest measured vancomycin and tobramycin concentrations in periprosthetic fluid samples will be recorded for each participant during the study period. Cmax will be compared between the two study arms.
Any postoperative complication (non-infectious) | Perioperative/Periprocedural
  Complications including seroma requiring aspiration, hematoma, skin necrosis, dehiscence, or unplanned return to the operating room within 90 days will be documented and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ara A Salibian, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the inclusion of sensitive health information and standardized photographs that cannot be fully de-identified. Data will be used solely for the purposes of this study in accordance with UC Davis IRB approval.